CLINICAL TRIAL: NCT04279977
Title: Impact of Initial Stroke Rehabilitation Placement on Functional Recovery and Cost-effectiveness
Brief Title: Stroke Rehabilitation, Functional Recovery, and Cost-effectiveness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Heather Hayes, Assistant Professor, University of Utah
Other Study IDs: 1K01HD097280-01 (NIH)
Record Dates: First submitted 2019-11-22; First posted 2020-02-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: rehabilitation; discharge; inpatient rehabilitation; skilled nursing; activity measure for post-acute care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatient Rehabilitation Facility: Individuals post-stroke who are discharged to an inpatient rehabilitation facility.
- Skilled Nursing Facility: Individuals post-stroke who are discharged to a skilled nursing facility.

SUMMARY:
The investigators will determine the client and non-client variables associated with discharge to an inpatient rehabilitation facility vs. skilled nursing facility in individuals' post-stroke. The investigators will determine how these variables are associated with short-term (discharge from facility) and long-term (6-months post-stroke) function and quality of life.

DETAILED DESCRIPTION:
This is a K01 award application for Dr. Heather Hayes, a neurologic rehabilitation therapist and a young investigator pursuing rehabilitation health services research to optimize post-acute rehabilitation care for patients after stroke. A K01 award will provide Dr. Hayes with the means to acquire critical skills in three key career development areas: 1) health services and policy research, 2) comparative effectiveness and outcomes research, and 3) cost-effective analyses. By acquiring these skills, Dr. Hayes will fulfill the career goal of becoming an independent rehabilitation scientist in health services research. To pursue this goal, Dr. Hayes has assembled an exceptional mentoring team complemented by a strong statistical advisor and proposes strong research aims that provide experiential learning in support of the career development objectives.

Stroke is a leading cause of long-term disability in the United States. A large portion of the cost of stroke care is rehabilitation. Providing optimal rehabilitation services aids in mitigating long-term disability for people after stroke. There are a lack of clinical guidelines and poor understanding of long-term outcomes after discharge from acute care to an inpatient rehabilitation facility (IRF) or skilled nursing facility (SNF) for individuals poststroke. The current healthcare climate requires faster decision making and early discharge, and the results may be inappropriate discharge to an IRF or SNF, and thus not providing the patient with optimal outcomes. By completing the following specific aims, the applicant aims to inform clinicians in the acute care setting about discharge placement and which rehabilitation service will lead to optimal individual and cost-effective outcomes after stroke. Specific Aim 1 will determine client (e.g., stroke severity, co-morbidities, and sociodemographic) and non-client (e.g., bed availability and insurance) variables identified at the end of the acute hospital stay to determine which of these variables are associated with discharge to an IRF or SNF. Specific Aim 2 will follow the clients to determine which of these client and non-client variables are associated with functional change- based on the Activity Measure for Post-Acute Care (AM-PAC) Inpatient "6-Clicks" Basic Mobility, Daily Activity, and Applied Cognitive tools at short-term (after discharge from IRF or SNF) and long-term (6-months poststroke). Specific Aim 3 will identify cost-effective strategies of placement into an IRF, to a SNF, and a tailored approach to IRF vs. SNF placement, based on client characteristics. Markov modeling will be used to predict related costs and quality-adjusted life years using the Health-Related Quality of Life in Stroke Patients.

Understanding the outcomes within these similar post-acute care settings (IRF/SNF) for stroke is important in a rapidly evolving healthcare climate. This study is significant because it will provide data about what initial client and non-client variables predict long-term outcomes after discharge to an IRF or SNF and identify cost-effective strategies based on these variables.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 years of age
* acute ischemic stroke

Exclusion Criteria:

* hemorrhagic stroke
* prior living status was at a long-term care facility.
* Transient ischemic attack
* being discharged to home, home with rehab or long term care
* not able to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Activity Measure for Post-Acute Care, Basic Mobility, change over time | baseline (acute care hospital stay) to discharge from IRF / SNF or 60 days max
  The Activity Measure for Post-Acute Care (AM-PAC) "6 Clicks" tools are comprised of six questions. Answers are based on a 4-point Likert scale ranging from 1-unable or total assistance to 4-no assistance or no difficulty. Scores range from 6 to 24, with lower scores indicating more assistance is required. The AM-PAC has a high degree of consistency between proxy (clinician or family) and client self-report in clients with stroke and has good reliability (ICC = 0.85) and validity (internal consistency = 0.96). The AM-PAC Basic Mobility domain assesses turning over in bed, sitting down and standing up, getting out of bed, transferring, walking, and stair climbing.
Activity Measure for Post-Acute Care, Daily Activity | baseline (acute care hospital stay) to discharge from IRF / SNF or 60 days max
  The AM-PAC Daily Activity domain assesses putting on and off clothing, bathing, toileting, grooming, and eating.Answers are based on a 4-point Likert scale ranging from 1-unable or total assistance to 4-no assistance or no difficulty. Scores range from 6 to 24, with lower scores indicating more assistance is required. The AM-PAC has a high degree of consistency between proxy (clinician or family) and client self-report in clients with stroke and has good reliability (ICC = 0.85) and validity (internal consistency = 0.96).
Activity Measure for Post-Acute Care, Applied Cognition | baseline (acute care hospital stay) to discharge from IRF / SNF or 60 days max
  The AM-PAC Applied Cognitive domain assesses comprehension and memory.Answers are based on a 4-point Likert scale ranging from 1-unable or total assistance to 4-no assistance or no difficulty. Scores range from 6 to 24, with lower scores indicating more assistance is required. The AM-PAC has a high degree of consistency between proxy (clinician or family) and client self-report in clients with stroke and has good reliability (ICC = 0.85) and validity (internal consistency = 0.96). .
Determination of client and non-client variables associated with discharge to an IRF / SNF | discharge from acute hospital stay or 20 days max.
  Client variables will include modified Rankin Scale, Stroke classification, hemiparetic side, presence of neglect, stroke severity, body mass index, comprehensive severity index, length of stay, co-morbidities, depression, age, gender, race, ethnicity, education, socioeconomic status, marital status, family / caregiver support. Non-client variables will include bed availability in facility, insurance, home set up, client / family preference, geographical location to facility and home.
Identify cost-effective strategies for IRF / SNF placement after stroke based on client and non-client variables. | Information will be collected on HRQOLSP at 6 months post-stroke.
  Evaluate the cost-effectiveness of three care strategies after stroke; 1) IRF placement; 2) SNF placement; and 3) tailored approach to an IRF vs. SNF placement, based on client characteristics. We will capture health related quality of life in stroke (HRQOLSP) patients to predict quality-adjusted life years and related costs.
Identify cost-effective strategies for IRF / SNF placement after stroke based on client and non-client variables. | Information will be collected on EQ-5D at 6 months post-stroke.
  Evaluate the cost-effectiveness of three care strategies after stroke; 1) IRF placement; 2) SNF placement; and 3) tailored approach to an IRF vs. SNF placement, based on client characteristics. We will capture EQ-5D to predict quality-adjusted life years and related costs.

SECONDARY OUTCOMES:
Activity Measure for Post-Acute Care, Basic Mobility, change over time | baseline (acute care hospital stay) to 6 months post-stroke
  The Activity Measure for Post-Acute Care (AM-PAC) "6 Clicks" tools are comprised of six questions. Answers are based on a 4-point Likert scale ranging from 1-unable or total assistance to 4-no assistance or no difficulty. Scores range from 6 to 24, with lower scores indicating more assistance is required. The AM-PAC has a high degree of consistency between proxy (clinician or family) and client self-report in clients with stroke and has good reliability (ICC = 0.85) and validity (internal consistency = 0.96). The AM-PAC Basic Mobility domain assesses turning over in bed, sitting down and standing up, getting out of bed, transferring, walking, and stair climbing.
Activity Measure for Post-Acute Care, Daily Activity | baseline (acute care hospital stay) to 6 months post-stroke
  The AM-PAC Daily Activity domain assesses putting on and off clothing, bathing, toileting, grooming, and eating.The Activity Measure for Post-Acute Care (AM-PAC) "6 Clicks" tools are comprised of six questions. Answers are based on a 4-point Likert scale ranging from 1-unable or total assistance to 4-no assistance or no difficulty. Scores range from 6 to 24, with lower scores indicating more assistance is required. The AM-PAC has a high degree of consistency between proxy (clinician or family) and client self-report in clients with stroke and has good reliability (ICC = 0.85) and validity (internal consistency = 0.96).
Activity Measure for Post-Acute Care, Applied Cognition | baseline (acute care hospital stay) to 6 months post-stroke
  The AM-PAC Applied Cognitive domain assesses comprehension and memory.The Activity Measure for Post-Acute Care (AM-PAC) "6 Clicks" tools are comprised of six questions. Answers are based on a 4-point Likert scale ranging from 1-unable or total assistance to 4-no assistance or no difficulty. Scores range from 6 to 24, with lower scores indicating more assistance is required. The AM-PAC has a high degree of consistency between proxy (clinician or family) and client self-report in clients with stroke and has good reliability (ICC = 0.85) and validity (internal consistency = 0.96).
Identify cost-effective strategies for IRF / SNF placement after stroke based on client and non-client variables. | Information will be collected on HRQOLSP at 12 months post-stroke.
  Evaluate the cost-effectiveness of three care strategies after stroke; 1) IRF placement; 2) SNF placement; and 3) tailored approach to an IRF vs. SNF placement, based on client characteristics. We will capture health related quality of life in stroke patients (HRQOLSP).
Identify cost-effective strategies for IRF / SNF placement after stroke based on client and non-client variables. | Information will be collected on EQ-5D at 6 months post-stroke.
  Evaluate the cost-effectiveness of three care strategies after stroke; 1) IRF placement; 2) SNF placement; and 3) tailored approach to an IRF vs. SNF placement, based on client characteristics. We will capture EQ-5D to predict quality-adjusted life years and related costs.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Hayes, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Looking into resources for where to store.